CLINICAL TRIAL: NCT06344247
Title: Comparison of the Efficacy and Safety of Sodium-glucose Cotransporter 2 Inhibitors and Glucagon-like Peptide-1 Receptor Agonists in Obese Patients With Kidney Disease: a Single Center, Prospective, Exploratory Study
Brief Title: Comparison of the Efficacy and Safety of SGLT2i and GLP-1 Receptor Agonists in Obese Patients With Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-0253
Record Dates: First submitted 2024-03-17; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Chronic Kidney Diseases
Keywords: Obesity; Chronic kidney disease; Sodium glucose cotransporter 2 inhibitors (SGLT2i); Glucagon like peptide-1 receptor agonists (GLP-1RA)
MeSH Terms: conditions — Obesity; Renal Insufficiency, Chronic | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Basic treatment (Experimental): RAS inhibitors（Losartan®️/Valsartan®️） : maintain the maximum dose/maximum tolerated dose.
  Interventions: Drug: RAS inhibitors：Losartan®️/Valsartan®️
- Basic treatment+SGLT2i (Experimental): On the basis of RAS inhibitors treatment, combined with dapagliflozin and titrated to the target dose (10 mg qd).
  Interventions: Drug: RAS inhibitors：Losartan®️/Valsartan®️; Drug: dapagliflozin：Forxiga®️
- Basic treatment+GLP-1RA (Experimental): On the basis of RAS inhibitors treatment, combined with semaglutide titrated to the target dose (1 mg qw).
  Interventions: Drug: RAS inhibitors：Losartan®️/Valsartan®️; Drug: simagliptin：Forxiga®️
- Basic treatment+SGLT2i+GLP-1RA (Experimental): On the basis of RAS inhibitors treatment, combined with dapagliflozin titrated to the target dose (10 mg qd) and semaglutide titrated to the target dose (1 mg qw).
  Interventions: Drug: RAS inhibitors：Losartan®️/Valsartan®️; Drug: dapagliflozin：Forxiga®️; Drug: simagliptin：Forxiga®️

INTERVENTIONS:
Drug: RAS inhibitors：Losartan®️/Valsartan®️ — Losartan®️/Valsartan®️ : maintain the maximum dose/maximum tolerated dose.
Drug: dapagliflozin：Forxiga®️ — Forxiga®️ : titrated to the target dose (10 mg qd).
  Arms: Basic treatment+SGLT2i; Basic treatment+SGLT2i+GLP-1RA
Drug: simagliptin：Forxiga®️ — Semaglutide®️ : titrated to the target dose (1 mg qw).
  Other Names: Semaglutide®️
  Arms: Basic treatment+GLP-1RA; Basic treatment+SGLT2i+GLP-1RA

SUMMARY:
The goal of this clinical trial is to exploring the changes in 24-hour urinary protein and renal function in obese patients with kidney disease after the application of sodium glucose cotransporter 2 inhibitors (SGLT2i) and glucagon like peptide-1 receptor agonists (GLP-1RA).

Eligible patients were randomly and non-blindly allocated to four groups in a 1:1:1:1 ratio.The first group is the optimized treatment group, and patients in this group maintain the maximum dose/maximum tolerated dose of RAS blocker therapy.

The second group is the optimized treatment + SGLT2i group. Participants in this group are titrated to the target dose (10 mg qd) in combination with dapagliflozin on the basis of optimized treatment.

The third group is the optimized treatment + GLP-1RA group. Participants in this group will be titrated to the target dose (1mg qw) in combination with semaglutide on the basis of optimized treatment.

The last group is the optimized treatment + SGLT2i + GLP-1RA treatment group, that is, based on the optimized treatment, combined with dapagliflozin titrated to the target dose (10 mg qd) and semaglutide titrated to the target dose (1 mg qw).

ELIGIBILITY:
Inclusion Criteria:

1. Agree to join this study and sign an informed consent form;
2. Age ≥ 18 years old and<75 years old;
3. BMI ≥ 25kg/m ² Or waist circumference ≥ 85cm (male)/≥ 80cm (female) or waist to hip ratio ≥ 0.9 (male)/≥ 0.85 (female);
4. Confirmed obesity related kidney disease through renal biopsy within six months;
5. Have received optimized treatment with RAS blockers and/or MRA for at least 3 months;

Exclusion Criteria:

1. Diagnosed as secondary obesity, such as hypothyroidism, Cushing's syndrome, polycystic ovary syndrome, etc;
2. Severe renal insufficiency (renal function eGFR<25 ml/min/1.73m2);
3. There is acute kidney injury; Defined as: (1) An increase in blood creatinine of ≥ 26.5 within 48 hours μ Mol/L; (2) Within 7 days, the increase in blood creatinine exceeds 1.5 times the baseline value or more; (3) Reduced urine output (<0.5 ml/kg/h) and lasting for more than 6 hours.
4. Symptoms of active reproductive and urinary system infections
5. Severe liver dysfunction (ALT/AST greater than 2.5 times the upper normal limit);
6. Severe cardiovascular and cerebrovascular diseases, rheumatic and immune diseases;
7. Serious metabolic diseases, such as diabetes ketoacidosis, hypertonic hyperglycemia, etc;
8. Late stage malignant tumors;
9. Have a known history of using drugs that affect glucose and lipid metabolism, such as glucocorticoids, antibiotics, anti anxiety or antidepressants, etc;
10. Severe bleeding tendency and inability to complete venous blood collection;
11. There are contraindications for MRI examination, such as patients with pacemakers, nerve stimulators, artificial metal heart valves, etc; Patients with claustrophobia; Epilepsy patients, etc.
12. Pregnant/lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of 24-hour urine protein quantification | 4、12、24、36、48 WEEK
  According to KDIGO 2021 glomerular disease management guidelines. ① Remission: proteinuria is reduced, and serum albumin is >30g/L. Renal function is stable. Complete remission (CR): proteinuria is significantly reduced, 24HUTP<0.3g/L, and serum albumin>30g/L. Renal function is stable. Partial response (PR): proteinuria decreases, 24HUTP decreases >50% from baseline and >0.3g/L. Serum albumin>30g/L. Renal function is stable.
  ② Invalid: proteinuria is not reduced compared with baseline, and serum albumin is <30g/L. Renal function is stable or declining.
  ③Relapse: After achieving CR or PR, proteinuria increases (24-hour urine protein quantification ≥3.5g/d) and serum albumin decreases, <30g/L. Renal function is stable or declining.

SECONDARY OUTCOMES:
Decline in glomerular filtration rate | 4、12、24、36、48 WEEK
Changes in BMI | 4、12、24、36、48 WEEK
  Body mass index
changes in fasting blood glucose | 4、12、24、36、48 WEEK

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai JIAO TONG University school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No